CLINICAL TRIAL: NCT01854931
Title: Translating an Effective Fall Prevention Program Into a Community-Based Practice
Brief Title: Community Dissemination of Tai Ji Quan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AG034956-02
Record Dates: First submitted 2013-05-09; First posted 2013-05-16 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Older Adults at Risk of Falling
Keywords: Tai Ji Quan; fall prevention; community dissemination
MeSH Terms: interventions — Tai Ji

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tai Ji Quan (Other): Single aim intervention - 2 twice per week for 48 weeks
  Interventions: Behavioral: Tai Ji Quan

INTERVENTIONS:
Behavioral: Tai Ji Quan — single aim intervention

SUMMARY:
The overarching objective of this project is to assess the potential public health impact of delivering Tai Ji Quan: Moving for Better Balance, a proven fall prevention program, through local community dissemination partners (e.g., senior service providers), in the selected counties in the state of Oregon.

DETAILED DESCRIPTION:
The program, Tai Chi: Moving for Better Balance, developed by ORI scientists (2003; 2004; 2008, a,b) was implemented in this dissemination project. Class duration was 90 minutes, 2-times per week over a 12-month period. During the initial 2 weeks, practice involved learning and performing 2 forms practiced in one set of 8 repetitions (for each form) and increased to a set of 10 repetitions for up to 5 forms between Week 3 and Week 5. Although additional forms were learned as the intervention progressed, starting in Week 6, training focused on 10-12 repetitions of the combination of forms rather than single forms. Once all 8 forms were learned ( Week 10), training was maintained at between 10-15 repetitions of the 8-form routine. Exercise activities were accompanied by music. Each Tai Chi practice session included (a) a 10-15 minute warm-up, (b) 60 minutes of Tai Chi practice, and (c) a 10-minute cool-down period. Instruction comprised (a) learning new movements and (b) reviewing movements learned from previous sessions. In addition, copies of the videotape/DVD and user's guidebook were distributed to all participants who were encouraged to use these materials for additional home practice.

All participating individuals were assessed at baseline, 6 months (mid-point), 12 months (intervention termination), and 6 months following the intervention (post-intervention follow-up) on measures of health, fall history, functional ability, and quality-of-life. Each evaluation session lasted about one hour and was conducted by a trained research assessor in various centers where these classes were held.

ELIGIBILITY:
Inclusion Criteria:

(a) 65 years of age or over, (b) physically mobile (i.e., can walk one or two blocks with or without an assistive device), and (c) medical clearance by a healthcare provider.

Exclusion Criteria:

(a) severe cognitive deficits defined by Mini-Mental State Evaluation, and (b) unable to commit for the 12 month duration of the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 511 (Actual)
Dates: Start 2012-05; Primary Completion 2016-12 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
adoption - defined as community centers that agree to participate (from the total number of centers approached within the dissemination geographic area) | at the study entry
  Target senior centers will be contacted to determine the willingness to adopt the program.

SECONDARY OUTCOMES:
Reach - defined by the total number of older adults agreed to participate | study on-set
  This indicator will be determined at the study on-set by documenting number of individuals who express interest in participating and are eventually enrolled in the program.

OTHER OUTCOMES:
implementation, effectiveness, maintenance | 12 months evaluation on program implementation and effectiveness, and a follow-up at month 18 on program maintenance
  Assessment of implementation includes fidelity evaluation (compliance rate, completion of required teaching and practice protocol).
  Effectiveness will be evaluated using falls calendar, physical performance based measures including Functional Reach, Timed Up&Go, 50 foot walk for speed.
  Maintenance will be evaluated by measuring continued participation among participants (individual level) and participating centers' (center level) willingness to continue the program.

CONTACTS AND LOCATIONS:
Overall Officials: Fuzhong Li, Ph.D., Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States

REFERENCES:
- [Derived] Li F, Harmer P, Fitzgerald K. Implementing an Evidence-Based Fall Prevention Intervention in Community Senior Centers. Am J Public Health. 2016 Nov;106(11):2026-2031. doi: 10.2105/AJPH.2016.303386. Epub 2016 Sep 15. PMID 27631751
- [Derived] Li F, Harmer P. Protocol for disseminating an evidence-based fall prevention program in community senior centers: evaluation of translatability and public health impact via a single group pre-post study. Implement Sci. 2014 May 26;9:63. doi: 10.1186/1748-5908-9-63. PMID 24884784